CLINICAL TRIAL: NCT02438722
Title: A Randomized Phase II/III Trial of Afatinib Plus Cetuximab Versus Afatinib Alone in Treatment-Naive Patients With Advanced, EGFR Mutation Positive Non-small Cell Lung Cancer (NSCLC)
Brief Title: S1403, Afatinib Dimaleate With or Without Cetuximab in Treating Patients With Newly Diagnosed Stage IV or Recurrent, EGFR Mutation Positive Non-small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S1403; NCI-2014-02405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); BI 1200.124; S1403 (Other: SWOG); S1403 (Other: CTEP); U10CA180888 (NIH)
Record Dates: First submitted 2015-05-06; First posted 2015-05-08 (Estimated); Results first posted 2021-03-17 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (afatinib dimaleate, cetuximab) (Experimental): Patients receive afatinib dimaleate PO QD on days 1-28 and cetuximab IV over 2 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Afatinib Dimaleate; Biological: Cetuximab; Other: Laboratory Biomarker Analysis
- Arm II (afatinib dimaleate) (Active Comparator): Patients receive afatinib dimaleate as in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Afatinib Dimaleate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Afatinib Dimaleate — Given PO
  Other Names: (2E)-N-(4-((3-Chloro-4-fluorophenyl)amino)-7-(((3S)-tetrahydrofuran-3-yl)oxy)quinazolin- 6-yl)-4-(dimethylamino)but-2-enamide bis(hydrogen (2Z)-but-2-enedioate); BIBW 2992MA2; BIBW2992 MA2; Gilotrif
Biological: Cetuximab — Given IV
  Other Names: Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
  Arms: Arm I (afatinib dimaleate, cetuximab)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II/III trial studies how well afatinib dimaleate with cetuximab works and compares it with afatinib dimaleate alone in treating patients with newly diagnosed stage IV or recurrent (has come back), epidermal growth factor receptor (EGFR) mutation positive non-small cell lung cancer. Afatinib dimaleate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, may block tumor growth in different ways by targeting certain cells. It is not yet known whether afatinib dimaleate is more effective when given alone or with cetuximab in treating patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if there is sufficient evidence to continue to the phase III component by comparing progression-free survival (PFS) between patients randomized to afatinib (afatinib dimaleate) in combination with cetuximab versus afatinib alone in the first-line treatment of patients with advanced EGFR-mutant non-small cell lung cancer (NSCLC). (Phase II) II. To determine the efficacy of the combination of afatinib and cetuximab compared to afatinib alone as measured by overall survival (OS) in the first-line treatment of patients with advanced EGFR-mutant NSCLC. (Phase III)

SECONDARY OBJECTIVES:

I. To evaluate the overall response rate (confirmed and unconfirmed, complete and partial responses) in the subset of patients with measurable disease treated with afatinib plus cetuximab compared to afatinib alone.

II. To assess the safety of each treatment arm when used in the first-line setting.

III. To compare time to treatment failure and time to treatment discontinuation between randomized to afatinib in combination with cetuximab versus afatinib alone.

TERTIARY OBJECTIVES:

I. To investigate the molecular mechanisms that confer benefit from afatinib and afatinib plus cetuximab by evaluating whether the presence of de novo EGFR T790M mutation or other molecular alterations in the pre-treatment tumor influence the clinical outcomes.

II. To quantitatively assess whether the ratio of sensitizing EGFR (EGFRs) mutation to EGFR T790M influences outcome and is altered during treatment.

III. To evaluate the frequency of known mechanisms of resistance to EGFR-directed therapies in the context of afatinib plus cetuximab and afatinib alone treatment.

IV. To identify potential novel predictors of benefit to afatinib plus cetuximab.

V. To identify potential new mechanisms of resistance to EGFR-directed therapies.

VI. To establish patient-derived xenografts (PDXs) from a subset of patients by re-biopsy at the time of progressive disease for drug testing and genomic analysis.

VII. To assess whether circulating tumor markers can be used as indicators of sensitivity and resistance to afatinib plus cetuximab and afatinib alone.

VIII. To determine whether the levels of EGFR protein by immunohistochemistry predict for benefit to afatinib plus cetuximab and afatinib alone.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive afatinib dimaleate orally (PO) once daily (QD) on days 1-28 and cetuximab intravenously (IV) over 2 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive afatinib dimaleate as in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed stage IV (American Joint Committee on Cancer [AJCC] 7th Edition) or recurrent non-small cell lung cancer (NSCLC)
* Patients must have documented presence of an EGFR exon 19 deltion or exon 21 (L858R) substitution mutation; T790M mutation or other molecular abnormality will be allowed as long as it accompanies one of the mutations listed above; EGFR testing must be performed using a Food and Drug Administration (FDA)-approved test or in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
* Patients must have tissue available and must agree to submission of tissue and blood; one to two paraffin-embedded tissue blocks or 15-20 unstained slides are requested (a minimum of 12 slides is required); cytology (i.e. fine-needle aspirations, pleural effusion specimens) is acceptable if a cell block or sufficient unstained slides are available; tumor material must be reviewed by a local pathologist who must confirm that at least 100 viable tumor cells are present in the sample and sign the S1403 Pathology Review Form; patients must also be willing to submit blood samples for correlative research at baseline, during treatment and at progression
* Patients enrolled at sites participating in the Repeat Biopsy Study must agree to submission of tissue obtained by a repeat biopsy performed at the time of disease progression
* Patients must not have received any prior systemic anticancer therapy for advanced or metastatic disease including chemotherapy or EGFR tyrosine kinase inhibitor therapy (including gefitinib, erlotinib, afatinib, or any experimental EGFR tyrosine kinase inhibitors [TKI] agents); prior chemotherapy for non-metastatic disease (i.e. adjuvant therapy or concurrent chemo-radiotherapy) is allowed as long as > 12 months has passed since completion of therapy; adjuvant EGFR-directed therapy is not allowed; local therapy (i.e. palliative radiotherapy) is allowed as long as a period of 7 days has passed since the last dose was received and the patient has recovered from any associated toxicity at the time of registration
* Patients may have measurable or non-measurable disease documented by computed tomography (CT) or magnetic resonance imaging (MRI) within 42 days prior to registration; the CT from a combined positron emission tomography (PET)/CT may be used only if it is of diagnostic quality; laboratory parameters are not acceptable as the only evidence of disease; in order to qualify as measurable, measurable disease must be outside previous radiation field; all disease must be assessed and documented on the Baseline Tumor Assessment Form (Response Evaluation Criteria in Solid Tumors [RECIST] 1.1)
* Patients must have a CT or MRI scan of the brain to evaluate for central nervous system (CNS) disease within 42 days prior to registration; patient must not have symptomatic brain metastases or evidence of leptomeningeal carcinomatosis; patients with asymptomatic brain metastases are eligible if off of steroids for at least 7 days prior to registration without development of symptoms
* Patients must not have any known clinically active interstitial lung disease
* Absolute neutrophil count (ANC) >= 1,500/mcL
* Platelets >= 75,000/mcL
* Hemoglobin >= 9 g/dL
* Total bilirubin =< 1.5 x institutional upper limit of normal (IULN)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x IULN (or =< 5 x IULN for patients with known liver metastases)
* Serum creatinine =< 1.5 x IULN OR measured or calculated creatinine clearance >= 60 mL/min
* Patients must not have significant gastrointestinal disorders with diarrhea as a major symptom (e.g. Crohn's disease, malabsorption, etc)
* Patients must be able to swallow medication by oral route
* Patients must not have a history of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure New York Heart Association (NYHA) classification of 3, unstable angina or poorly controlled arrhythmia or myocardial infarction within 6 months prior to registration; if clinically indicated, echocardiogram or multigated acquisition (MUGA) must be performed and cardiac ejection fraction must be >= 50%
* Patients must not have had major surgery within 28 days prior to registration or be scheduled for surgery during the projected course of protocol treatment; tumor biopsy is allowed
* Patients must not have a known history of active hepatitis B infection (defined as presence of hepatitis B surface antigen [Hep B sAg] and/ or Hep B deoxyribonucleic acid [DNA]), active hepatitis C infection (defined as presence of hepatitis C [Hep C] ribonucleic acid [RNA]) and/or known human immunodeficiency virus (HIV) seropositive
* Patients must not have any other concomitant serious illness or organ system dysfunction which in the opinion of the investigator would either compromise patient safety or interfere with the evaluation of the safety of the study drug
* Patients must not be planning to receive any other investigational agents during the course of protocol treatment
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to afatinib and/or cetuximab
* Prestudy history and physical must be obtained with 28 days prior to registration
* Patients must have Zubrod performance status of 0 - 2
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease free for three years
* Patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method; a woman is considered to be of "reproductive potential" if she has had menses at any time in the preceding 12 consecutive months; in addition to routine contraceptive methods, "effective contraception" also includes heterosexual celibacy and surgery intended to prevent pregnancy (or with a side-effect of pregnancy prevention) defined as a hysterectomy, bilateral oophorectomy or bilateral tubal ligation; however, if at any point a previously celibate patient chooses to become heterosexually active during the time period for use of contraceptive measures outlined in the protocol, he/she is responsible for beginning contraceptive measures
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* As a part of the Oncology Patient Enrollment Network (OPEN) registration process the treating institution's identity is provided in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered in the system

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2015-05-07 (Actual); Primary Completion 2018-09-25 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Goldberg, Principal Investigator — SWOG Cancer Research Network
Locations (638):
- United States (638):
  - Mercy Hospital Fort Smith, Fort Smith, Arkansas
  - CHI Saint Vincent Cancer Center Hot Springs, Hot Springs, Arkansas
  - Fowler Family Center for Cancer Care, Jonesboro, Arkansas
  - Kaiser Permanente-Anaheim, Anaheim, California
  - PCR Oncology, Arroyo Grande, California
  - Sutter Auburn Faith Hospital, Auburn, California
  - Sutter Cancer Centers Radiation Oncology Services-Auburn, Auburn, California
  - AIS Cancer Center at San Joaquin Community Hospital, Bakersfield, California
  - Kaiser Permanente-Baldwin Park, Baldwin Park, California
  - Kaiser Permanente-Bellflower, Bellflower, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills-Peninsula Medical Center, Burlingame, California
  - Sutter Cancer Centers Radiation Oncology Services-Cameron Park, Cameron Park, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Sutter Davis Hospital, Davis, California
  - Kaiser Permanente-Fontana, Fontana, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Kaiser Permanente - Harbor City, Harbor City, California
  - Kaiser Permanente-Irvine, Irvine, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Kaiser Permanente-Cadillac, Los Angeles, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Mercy UC Davis Cancer Center, Merced, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Cancer Centers Radiation Oncology Services-Roseville, Roseville, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Kaiser Permanente-San Diego Mission, San Diego, California
  - Kaiser Permanente-San Diego Zion, San Diego, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Kaiser Permanente-San Marcos, San Marcos, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Sutter Pacific Medical Foundation, Santa Rosa, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Gene Upshaw Memorial Tahoe Forest Cancer Center, Truckee, California
  - Northbay Cancer Center, Vacaville, California
  - Sutter Cancer Centers Radiation Oncology Services-Vacaville, Vacaville, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Kaiser Permanente-Woodland Hills, Woodland Hills, California
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers-Penrose, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Mercy Medical Center, Durango, Colorado
  - Southwest Oncology PC, Durango, Colorado
  - Mountain Blue Cancer Care Center, Golden, Colorado
  - Rocky Mountain Cancer Centers-Lakewood, Lakewood, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Littleton Adventist Hospital, Littleton, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - Rocky Mountain Cancer Centers-Longmont, Longmont, Colorado
  - Parker Adventist Hospital, Parker, Colorado
  - Rocky Mountain Cancer Centers-Parker, Parker, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - Rocky Mountain Cancer Centers - Pueblo, Pueblo, Colorado
  - Rocky Mountain Cancer Centers-Thornton, Thornton, Colorado
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Yale-New Haven Shoreline Medical Center, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Smilow Cancer Hospital-Orange Care Center, Orange, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Delaware Clinical and Laboratory Physicians PA, Newark, Delaware
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Regional Hematology and Oncology PA, Newark, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Beebe Health Campus, Rehoboth Beach, Delaware
  - Nanticoke Memorial Hospital, Seaford, Delaware
  - Christiana Care Health System-Wilmington Hospital, Wilmington, Delaware
  - Baptist MD Anderson Cancer Center, Jacksonville, Florida
  - Sacred Heart Hospital, Pensacola, Florida
  - Central Georgia Gynecologic Oncology, Macon, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Memorial University Medical Center, Savannah, Georgia
  - Summit Cancer Care-Memorial, Savannah, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Low Country Cancer Care Associates PC, Savannah, Georgia
  - Summit Cancer Care-Candler, Savannah, Georgia
  - South Georgia Medical Center/Pearlman Cancer Center, Valdosta, Georgia
  - Hawaii Cancer Care Inc-POB II, Honolulu, Hawaii
  - Hawaii Oncology Inc-POB I, Honolulu, Hawaii
  - Island Urology, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - Hawaii Cancer Care Inc-Liliha, Honolulu, Hawaii
  - Hawaii Oncology Inc-Kuakini, Honolulu, Hawaii
  - Kuakini Medical Center, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Wilcox Memorial Hospital and Kauai Medical Clinic, Lihue, Hawaii
  - Hawaii Oncology Inc-Pali Momi, ‘Aiea, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - The Cancer Center of Hawaii-Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Medical Center, Coeur d'Alene, Idaho
  - Walter Knox Memorial Hospital, Emmett, Idaho
  - Idaho Urologic Institute-Meridian, Meridian, Idaho
  - Saint Alphonsus Medical Center-Nampa, Nampa, Idaho
  - Kootenai Cancer Center, Post Falls, Idaho
  - Kootenai Cancer Clinic, Sandpoint, Idaho
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Illinois CancerCare-Bloomington, Bloomington, Illinois
  - Illinois CancerCare-Canton, Canton, Illinois
  - Memorial Hospital of Carbondale, Carbondale, Illinois
  - SIH Cancer Institute, Carterville, Illinois
  - Illinois CancerCare-Carthage, Carthage, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Carle on Vermilion, Danville, Illinois
  - Cancer Care Specialists of Central Illinois, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Illinois CancerCare-Eureka, Eureka, Illinois
  - Illinois CancerCare-Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Illinois CancerCare-Kewanee Clinic, Kewanee, Illinois
  - Illinois CancerCare-Macomb, Macomb, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Spector, David MD (UIA Investigator), Moline, Illinois
  - Trinity Medical Center, Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Radiation Oncology of Northern Illinois, Ottawa, Illinois
  - Illinois CancerCare-Pekin, Pekin, Illinois
  - OSF Saint Francis Radiation Oncology at Pekin Cancer Treatment Center, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - OSF Saint Francis Radiation Oncology at Peoria Cancer Center, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois CancerCare-Peru, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Edward Hospital/Cancer Center?Plainfield, Plainfield, Illinois
  - Illinois CancerCare-Princeton, Princeton, Illinois
  - SwedishAmerican Regional Cancer Center/ACT, Rockford, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Cancer Care Specialists of Illinois-Swansea, Swansea, Illinois
  - Memorial and Saint Elizabeth's Health Care Services LLP, Swansea, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - Deaconess Clinic Downtown, Evansville, Indiana
  - Parkview Hospital Randallia, Fort Wayne, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Woodland Cancer Care Center, Michigan City, Indiana
  - Chancellor Center for Oncology, Newburgh, Indiana
  - Reid Health, Richmond, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - McFarland Clinic PC-Boone, Boone, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Mercy Cancer Center-West Lakes, Clive, Iowa
  - Alegent Health Mercy Hospital, Council Bluffs, Iowa
  - Greater Regional Medical Center, Creston, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - McFarland Clinic PC-Trinity Cancer Center, Fort Dodge, Iowa
  - McFarland Clinic PC-Jefferson, Jefferson, Iowa
  - McFarland Clinic PC-Marshalltown, Marshalltown, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Mercy Medical Center-West Lakes, West Des Moines, Iowa
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Coffeyville Regional Medical Center, Coffeyville, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Saint Catherine Hospital, Garden City, Kansas
  - Central Care Cancer Center - Great Bend, Great Bend, Kansas
  - Saint Rose Ambulatory and Surgery Center, Great Bend, Kansas
  - Hays Medical Center, Hays, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Cancer Center-West, Kansas City, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Kansas Institute of Medicine Cancer and Blood Center, Lenexa, Kansas
  - Minimally Invasive Surgery Hospital, Lenexa, Kansas
  - Cancer Center of Kansas-Liberal, Liberal, Kansas
  - Cancer Center of Kansas-Manhattan, Manhattan, Kansas
  - Cancer Center of Kansas - McPherson, McPherson, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Medical Center, Olathe, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - University of Kansas Cancer Center-Overland Park, Overland Park, Kansas
  - Saint Luke's South Hospital, Overland Park, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Via Christi Hospital-Pittsburg, Pittsburg, Kansas
  - Kansas City NCI Community Oncology Research Program, Prairie Village, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Saint Francis Hospital and Medical Center - Topeka, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Commonwealth Cancer Center-Corbin, Corbin, Kentucky
  - Oncology Hematology Care Inc-Crestview, Crestview Hills, Kentucky
  - Saint Joseph Radiation Oncology Resource Center, Lexington, Kentucky
  - Saint Joseph Hospital East, Lexington, Kentucky
  - Jewish Hospital, Louisville, Kentucky
  - Saints Mary and Elizabeth Hospital, Louisville, Kentucky
  - Jewish Hospital Medical Center Northeast, Louisville, Kentucky
  - Jewish Hospital Medical Center South, Shepherdsville, Kentucky
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - Lafayette Family Cancer Center-EMMC, Brewer, Maine
  - Penobscot Bay Medical Center, Rockport, Maine
  - Beverly Hospital, Beverly, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Addison Gilbert Hospital, Gloucester, Massachusetts
  - Winchester Hospital, Winchester, Massachusetts
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - IHA Hematology Oncology Consultants-Brighton, Brighton, Michigan
  - Saint Joseph Mercy Brighton, Brighton, Michigan
  - IHA Hematology Oncology Consultants-Canton, Canton, Michigan
  - Saint Joseph Mercy Canton, Canton, Michigan
  - Caro Cancer Center, Caro, Michigan
  - IHA Hematology Oncology Consultants-Chelsea, Chelsea, Michigan
  - Saint Joseph Mercy Chelsea, Chelsea, Michigan
  - Hematology Oncology Consultants-Clarkston, Clarkston, Michigan
  - Newland Medical Associates-Clarkston, Clarkston, Michigan
  - Beaumont Hospital-Dearborn, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Great Lakes Cancer Management Specialists-Doctors Park, East China Township, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Genesee Cancer and Blood Disease Treatment Center, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Great Lakes Cancer Management Specialists-Van Elslander Cancer Center, Grosse Pointe Woods, Michigan
  - Lymphoma Clinic of Michigan, Grosse Pointe Woods, Michigan
  - Michigan Breast Specialists-Grosse Pointe Woods, Grosse Pointe Woods, Michigan
  - Allegiance Health, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Hope Cancer Clinic, Livonia, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Medical Campus, Macomb, Michigan
  - Michigan Breast Specialists-Macomb Township, Macomb, Michigan
  - Saint Mary's Oncology/Hematology Associates of Marlette, Marlette, Michigan
  - UP Health System Hematology Oncology Marquette, Marquette, Michigan
  - UP Health System Marquette, Marquette, Michigan
  - Monroe Cancer Center, Monroe, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Lakeland Community Hospital, Niles, Michigan
  - 21st Century Oncology-Pontiac, Pontiac, Michigan
  - Hope Cancer Center, Pontiac, Michigan
  - Newland Medical Associates-Pontiac, Pontiac, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Huron Medical Center PC, Port Huron, Michigan
  - Lake Huron Medical Center, Port Huron, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Great Lakes Cancer Management Specialists-Rochester Hills, Rochester Hills, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Bhadresh Nayak MD PC-Sterling Heights, Sterling Heights, Michigan
  - Saint Joseph Health System-Tawas City, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Advanced Breast Care Center PLLC, Warren, Michigan
  - Bhadresh Nayak MD PC-Warren, Warren, Michigan
  - Great Lakes Cancer Management Specialists-Macomb Professional Building, Warren, Michigan
  - Macomb Hematology Oncology PC, Warren, Michigan
  - Michigan Breast Specialists-Warren, Warren, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Huron Gastroenterology PC, Ypsilanti, Michigan
  - IHA Hematology Oncology Consultants-Ann Arbor, Ypsilanti, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Fairview Maple Grove Medical Center, Maple Grove, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Health Partners Inc, Minneapolis, Minnesota
  - New Ulm Medical Center, New Ulm, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Lakeview Hospital, Stillwater, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - Fairview Lakes Medical Center, Wyoming, Minnesota
  - Baptist Memorial Hospital and Cancer Center-Union County, New Albany, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Oxford, Oxford, Mississippi
  - Singing River Hospital, Pascagoula, Mississippi
  - Baptist Memorial Hospital and Cancer Center-Desoto, Southhaven, Mississippi
  - Central Care Cancer Center - Bolivar, Bolivar, Missouri
  - Parkland Health Center-Bonne Terre, Bonne Terre, Missouri
  - Cox Cancer Center Branson, Branson, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Cancer Center, Cape Girardeau, Missouri
  - Centerpoint Medical Center LLC, Independence, Missouri
  - Capital Region Medical Center-Goldschmidt Cancer Center, Jefferson City, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital Joplin, Joplin, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Heartland Hematology and Oncology Associates Incorporated, Kansas City, Missouri
  - Kansas City Veterans Affairs Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-South, Kansas City, Missouri
  - Research Medical Center, Kansas City, Missouri
  - The University of Kansas Cancer Center-North, Kansas City, Missouri
  - The University of Kansas Cancer Center-Lee's Summit, Lee's Summit, Missouri
  - Saint Luke's East - Lee's Summit, Lee's Summit, Missouri
  - Liberty Radiation Oncology Center, Liberty, Missouri
  - Delbert Day Cancer Institute at PCRMC, Rolla, Missouri
  - Mercy Clinic-Rolla-Cancer and Hematology, Rolla, Missouri
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Sainte Genevieve County Memorial Hospital, Sainte Genevieve, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Missouri Baptist Sullivan Hospital, Sullivan, Missouri
  - Missouri Baptist Outpatient Center-Sunset Hills, Sunset Hills, Missouri
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Hospital, Missoula, Montana
  - CHI Health Saint Francis, Grand Island, Nebraska
  - Heartland Hematology and Oncology, Kearney, Nebraska
  - CHI Health Good Samaritan, Kearney, Nebraska
  - Nebraska Hematology and Oncology, Lincoln, Nebraska
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - Southeast Nebraska Cancer Center, Lincoln, Nebraska
  - Faith Regional Health Services Carson Cancer Center, Norfolk, Nebraska
  - Great Plains Health Callahan Cancer Center, North Platte, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Hematology and Oncology Consultants PC, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Nebraska Cancer Specialists - Omaha, Omaha, Nebraska
  - Alegent Health Lakeside Hospital, Omaha, Nebraska
  - Oncology Hematology West PC, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Midlands Community Hospital, Papillion, Nebraska
  - Regional West Medical Center Cancer Center, Scottsbluff, Nebraska
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Cancer and Blood Specialists-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada - Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Horizon Ridge, Henderson, Nevada
  - Las Vegas Cancer Center-Henderson, Henderson, Nevada
  - 21st Century Oncology-Henderson, Henderson, Nevada
  - Comprehensive Cancer Centers of Nevada-Southeast Henderson, Henderson, Nevada
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Cancer and Blood Specialists-Shadow, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Central, Las Vegas, Nevada
  - 21st Century Oncology, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Maryland Parkway, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-San Martin, Las Vegas, Nevada
  - Radiation Oncology Centers of Nevada Southeast, Las Vegas, Nevada
  - Cancer Therapy and Integrative Medicine, Las Vegas, Nevada
  - 21st Century Oncology-Vegas Tenaya, Las Vegas, Nevada
  - Ann M Wierman MD LTD, Las Vegas, Nevada
  - Cancer and Blood Specialists-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Northwest, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Tenaya, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada-Summerlin, Las Vegas, Nevada
  - Summerlin Hospital Medical Center, Las Vegas, Nevada
  - Las Vegas Cancer Center-Medical Center, Las Vegas, Nevada
  - 21st Century Oncology-Fort Apache, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Nevada Cancer Specialists-Fort Apache, Las Vegas, Nevada
  - HealthCare Partners Medical Group Oncology/Hematology-Centennial Hills, Las Vegas, Nevada
  - Comprehensive Cancer Centers of Nevada - Central Valley, Las Vegas, Nevada
  - University Cancer Center, Las Vegas, Nevada
  - Hope Cancer Care of Nevada-Pahrump, Pahrump, Nevada
  - Renown Regional Medical Center, Reno, Nevada
  - Saint Mary's Regional Medical Center, Reno, Nevada
  - Radiation Oncology Associates, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Norris Cotton Cancer Center-Manchester, Manchester, New Hampshire
  - Norris Cotton Cancer Center-Nashua, Nashua, New Hampshire
  - Englewood Hospital and Medical Center, Englewood, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Inspira Medical Center Vineland, Vineland, New Jersey
  - Inspira Medical Center Woodbury, Woodbury, New Jersey
  - Lovelace Medical Center-Saint Joseph Square, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - New Mexico Oncology Hematology Consultants, Albuquerque, New Mexico
  - Memorial Medical Center - Las Cruces, Las Cruces, New Mexico
  - Christus Saint Vincent Regional Cancer Center, Santa Fe, New Mexico
  - Orange Regional Medical Center, Middletown, New York
  - University of Rochester, Rochester, New York
  - Faxton-Saint Luke's Healthcare, Utica, New York
  - Cancer Care of Western North Carolina, Asheville, North Carolina
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Asheville Hematology-Oncology Associates, Asheville, North Carolina
  - Sampson Radiation Oncology, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Clinton, Clinton, North Carolina
  - Southeastern Medical Oncology Center-Goldsboro, Goldsboro, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Hendersonville Hematology and Oncology at Pardee, Hendersonville, North Carolina
  - Margaret R Pardee Memorial Hospital, Hendersonville, North Carolina
  - Park Ridge Hospital Breast Health Center, Hendersonville, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Southeastern Medical Oncology Center-Jacksonville, Jacksonville, North Carolina
  - Kinston Medical Specialists PA, Kinston, North Carolina
  - Southeastern Medical Oncology Center-Wilson, Wilson, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Roger Maris Cancer Center, Fargo, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Trinity Cancer Care Center, Minot, North Dakota
  - Akron General Medical Center, Akron, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Dayton Physicians LLC-Miami Valley South, Centerville, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Oncology Hematology Care Inc-Eden Park, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Mercy West, Cincinnati, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Oncology Hematology Care Inc - Anderson, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Kenwood, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - Oncology Hematology Care Inc-Blue Ash, Cincinnati, Ohio
  - TriHealth Cancer Institute-Westside, Cincinnati, Ohio
  - TriHealth Cancer Institute-Anderson, Cincinnati, Ohio
  - Columbus Oncology and Hematology Associates Inc, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Dayton Physicians LLC-Samaritan North, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Delaware Health Center-Grady Cancer Center, Delaware, Ohio
  - Delaware Radiation Oncology, Delaware, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Oncology Hematology Care Inc-Healthplex, Fairfield, Ohio
  - Armes Family Cancer Center, Findlay, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Orion Cancer Care, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Dayton Physicians LLC-Atrium, Franklin, Ohio
  - Dayton Physicians LLC-Wayne, Greenville, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Greater Dayton Cancer Center, Kettering, Ohio
  - First Dayton Cancer Care, Kettering, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Dayton Physicians LLC-Signal Point, Middletown, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Newark Radiation Oncology, Newark, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Dayton Physicians LLC-Wilson, Sidney, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Dayton Physicians LLC-Upper Valley, Troy, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Saint Alphonsus Medical Center-Baker City, Baker City, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Providence Medford Medical Center, Medford, Oregon
  - Rogue Valley Medical Center, Medford, Oregon
  - Saint Alphonsus Medical Center-Ontario, Ontario, Oregon
  - Kaiser Permanente Northwest, Portland, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - UPMC-Heritage Valley Health System Beaver, Beaver, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Christiana Care Health System-Concord Health Center, Chadds Ford, Pennsylvania
  - Ephrata Cancer Center, Ephrata, Pennsylvania
  - Ephrata Community Hospital, Ephrata, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Centers - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Cherry Tree Cancer Center, Hanover, Pennsylvania
  - UPMC-Johnstown/John P. Murtha Regional Cancer Center, Johnstown, Pennsylvania
  - Sechler Family Cancer Center, Lebanon, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - UPMC-Coraopolis/Heritage Valley Radiation Oncology, Moon Township, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC-Magee Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC-Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Margaret, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UPMC-Shadyside Hospital, Pittsburgh, Pennsylvania
  - UPMC-Passavant Hospital, Pittsburgh, Pennsylvania
  - UPMC-Saint Clair Hospital Cancer Center, Pittsburgh, Pennsylvania
  - Penn State Health Saint Joseph Medical Center, Reading, Pennsylvania
  - Guthrie Medical Group PC-Robert Packer Hospital, Sayre, Pennsylvania
  - UPMC Cancer Center at UPMC Northwest, Seneca, Pennsylvania
  - UPMC Uniontown Hospital Radiation Oncology, Uniontown, Pennsylvania
  - UPMC Washington Hospital Radiation Oncology, Washington, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - UPMC Susquehanna, Williamsport, Pennsylvania
  - WellSpan Health-York Cancer Center, York, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Greenville Health System Cancer Institute-Easley, Easley, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Saint Francis Hospital, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Butternut, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Faris, Greenville, South Carolina
  - Greenville Memorial Hospital, Greenville, South Carolina
  - Saint Francis Cancer Center, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Eastside, Greenville, South Carolina
  - Greenville Health System Cancer Institute-Greer, Greer, South Carolina
  - Greenville Health System Cancer Institute-Seneca, Seneca, South Carolina
  - Greenville Health System Cancer Institute-Spartanburg, Spartanburg, South Carolina
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Boston Baskin Cancer Center-Bartlett, Bartlett, Tennessee
  - Memorial Hospital, Chattanooga, Tennessee
  - Integrity Oncology PLLC-Collierville, Collierville, Tennessee
  - Vanderbilt-Ingram Cancer Center Cool Springs, Franklin, Tennessee
  - Pulmonary Medicine Center of Chattanooga-Hixson, Hixson, Tennessee
  - Baptist Memorial Hospital and Cancer Center-Memphis, Memphis, Tennessee
  - Baptist Memorial Hospital for Women, Memphis, Tennessee
  - Family Cancer Center-Memphis, Memphis, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Memorial GYN Plus, Ooltewah, Tennessee
  - Saint Joseph Regional Cancer Center, Bryan, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Norris Cotton Cancer Center-North, Saint Johnsbury, Vermont
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Harrison Medical Center, Bremerton, Washington
  - Highline Medical Center-Main Campus, Burien, Washington
  - Saint Elizabeth Hospital, Enumclaw, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Saint Clare Hospital, Lakewood, Washington
  - Harrison HealthPartners Hematology and Oncology-Poulsbo, Poulsbo, Washington
  - Franciscan Research Center-Northwest Medical Plaza, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Saint Mary's Medical Center, Huntington, West Virginia
  - Langlade Hospital and Cancer Center, Antigo, Wisconsin
  - Aurora Cancer Care-Southern Lakes VLCC, Burlington, Wisconsin
  - Marshfield Clinic-Chippewa Center, Chippewa Falls, Wisconsin
  - Marshfield Clinic Cancer Center - Eau Claire, Eau Claire, Wisconsin
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Health Center-Fond du Lac, Fond du Lac, Wisconsin
  - Aurora Health Care Germantown Health Center, Germantown, Wisconsin
  - Aurora Cancer Care-Grafton, Grafton, Wisconsin
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora Cancer Care-Kenosha South, Kenosha, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Marshfield Clinic - Ladysmith Center, Ladysmith, Wisconsin
  - Aurora Bay Area Medical Group-Marinette, Marinette, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Vince Lombardi Cancer Clinic-Marinette, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Marshfield Medical Center, Marshfield, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Aurora Cancer Care-Milwaukee, Milwaukee, Wisconsin
  - Columbia Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin
  - Aurora Sinai Medical Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - Vince Lombardi Cancer Clinic - Oshkosh, Oshkosh, Wisconsin
  - Aurora Cancer Care-Racine, Racine, Wisconsin
  - Lakeview Medical Center-Marshfield Clinic, Rice Lake, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Ascension Saint Michael's Hospital, Stevens Point, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Marshfield Clinic Stevens Point Center, Stevens Point, Wisconsin
  - Aurora Medical Center in Summit, Summit, Wisconsin
  - Vince Lombardi Cancer Clinic-Two Rivers, Two Rivers, Wisconsin
  - Aurora Cancer Care-Waukesha, Waukesha, Wisconsin
  - Aspirus Regional Cancer Center, Wausau, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Aurora Cancer Care-Milwaukee West, Wauwatosa, Wisconsin
  - Aurora West Allis Medical Center, West Allis, Wisconsin
  - Diagnostic and Treatment Center, Weston, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Aspirus UW Cancer Center, Wisconsin Rapids, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Big Horn Basin Cancer Center, Cody, Wyoming
  - Billings Clinic-Cody, Cody, Wyoming
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Derived] Goldberg SB, Redman MW, Lilenbaum R, Politi K, Stinchcombe TE, Horn L, Chen EH, Mashru SH, Gettinger SN, Melnick MA, Herbst RS, Baumgart MA, Miao J, Moon J, Kelly K, Gandara DR. Randomized Trial of Afatinib Plus Cetuximab Versus Afatinib Alone for First-Line Treatment of EGFR-Mutant Non-Small-Cell Lung Cancer: Final Results From SWOG S1403. J Clin Oncol. 2020 Dec 1;38(34):4076-4085. doi: 10.1200/JCO.20.01149. Epub 2020 Oct 6. PMID 33021871

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 174 participants were enrolled, however, 6 were deemed ineligible. Thus, 168 participants were eligible and randomized.
  5 participants on arm 1 did not receive protocol therapy.
Groups:
- Arm I (Afatinib Dimaleate, Cetuximab): Participants receive afatinib dimaleate PO QD on days 1-28 and cetuximab IV over 2 hours on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Afatinib Dimaleate: Given PO
  Cetuximab: Given IV
  Laboratory Biomarker Analysis: Correlative studies
- Arm II (Afatinib Dimaleate): Participants receive afatinib dimaleate as in Arm I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Afatinib Dimaleate: Given PO
  Laboratory Biomarker Analysis: Correlative studies
Period: Overall Study
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Started | 83 | 85
Participants Evaluable for Adverse Events | 78 | 85
Completed | 0 | 0
Not Completed | 83 | 85
Not completed — Adverse Event | 12 | 9
Not completed — Refusal unrelated to AE | 2 | 5
Not completed — Disease progression/relapse | 46 | 51
Not completed — Death | 0 | 3
Not completed — Physician Decision | 2 | 2
Not completed — Exceeded protocol-specified maximum treatment delay unrelated to AE | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — On protocol treatment | 15 | 14
Not completed — Did not receive protocol treatment | 5 | 0

BASELINE CHARACTERISTICS:
Population: Eligible participants that were randomized to study arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate) | Total
Number analyzed (Participants) | 83 | 85 | 168
Age, Continuous [Median (Full Range); unit: years] | 65.5 [27.9 to 90.5] | 66.3 [39.3 to 93.0] | 66.0 [27.9 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 53 | 112
  Male | 24 | 32 | 56
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 11 | 10 | 21
  Black | 3 | 8 | 11
  Multiracial | 1 | 0 | 1
  Native American | 2 | 0 | 2
  Pacific Islander | 0 | 1 | 1
  White | 59 | 63 | 122
  Unknown | 7 | 3 | 10
  Hispanic | 9 | 8 | 17
Performance status [Count of Participants; unit: Participants] — Participants were graded according to the Zubrod Performance Status Scale.
  0- Fully active, able to carry out on all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g. light housework, office work.
  2. Ambulatory and capable of self-care but unable to carry out any work activities; up and about more than 50% of waking hours.
  Participants
    0 | 38 | 32 | 70
    1 | 36 | 47 | 83
    2 | 9 | 6 | 15
EGFR mutation type [Count of Participants; unit: Participants]
  Exon 19 deletion | 53 | 54 | 107
  L858R mutation | 30 | 31 | 61
Histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 80 | 81 | 161
  Large cell | 0 | 1 | 1
  Squamous | 3 | 0 | 3
  Mixed (>= 50% squamous) | 0 | 1 | 1
  Mixed (< 50% squamous) | 0 | 1 | 1
  Other non-small cell | 0 | 1 | 1
Smoking history [Count of Participants; unit: Participants]
  Current smoker | 8 | 6 | 14
  Former smoker | 32 | 32 | 64
  Never smoker | 43 | 47 | 90
Weight loss in the last 6 months, % [Count of Participants; unit: Participants]
  <5 | 57 | 57 | 114
  5-10 | 13 | 15 | 28
  10-20 | 12 | 9 | 21
  >=20 | 0 | 1 | 1
  Data Missing | 1 | 3 | 4
Brain metastases [Count of Participants; unit: Participants] | 27 | 21 | 48

OUTCOME MEASURES:

1. Primary Outcome: 2-year Overall Survival Rate
Description: Percentage of participants still alive 2 years post registration.
  KM estimate at 2 years is presented, Overall Survival assessed for a total of 3 years in order to calculate value.
Time Frame: Up to 3 years post registration
Population: Eligible participants that were randomized to study arms.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Number analyzed (Participants) | 83 | 85
percentage of participants | 67 [55 to 76] | 70 [58 to 79]
Statistical Analysis 1: Comparison: Arm I (Afatinib Dimaleate, Cetuximab) vs Arm II (Afatinib Dimaleate); Test type: Superiority; p = 0.44, Log Rank; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.50 to 1.36]

2. Primary Outcome: Progression-Free Survival
Description: From date of registration to date of first documentation of progression or symptomatic deterioration or death due to any cause.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of appropriate diameters of target measurable lesions over smallest sum observed, as well as an absolute increase of at least 0.5 cm. Unequivocal progression of non-measurable disease in the opinion of treating physician. Appearance of any new lesion/site. Death due to disease without prior documentation of progression and without symptomatic deterioration.
Time Frame: up to 3 years post registration
Population: Eligible participants that were randomized to study arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Number analyzed (Participants) | 83 | 85
months | 11.9 [9.9 to 17.8] | 13.4 [9.3 to 14.9]
Statistical Analysis 1: Comparison: Arm I (Afatinib Dimaleate, Cetuximab) vs Arm II (Afatinib Dimaleate); Test type: Superiority; p = 0.94, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.72 to 1.43]

3. Secondary Outcome: Response Rates
Description: Percentage of participants with confirmed and unconfirmed, partial response and complete response to treatment Response Evaluation Criteria in Solid Tumors Criteria (RECIST 1.1).
  Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of appropriate diameters of all target measurable lesions; Overall Response (OR) = CR + PR.
Time Frame: Up to 3 years
Population: Eligible participants that were randomized to study arms and who had baseline measurable disease (153)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Number analyzed (Participants) | 76 | 77
percentage of participants | 67 [55 to 77] | 74 [63 to 83]

4. Secondary Outcome: Time to Treatment Discontinuation
Description: From date of registration to date of discontinuation of treatment or death due to any cause
Time Frame: up to 3 years post-registration
Population: Eligible participants who were randomized to study arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Number analyzed (Participants) | 83 | 85
months | 12.7 [10.8 to 17.6] | 12.2 [9.3 to 15.1]
Statistical Analysis 1: Comparison: Arm I (Afatinib Dimaleate, Cetuximab) vs Arm II (Afatinib Dimaleate); Test type: Superiority; p = 0.54, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.64 to 1.26]

5. Secondary Outcome: Time to Treatment Failure
Description: From date of registration to date of first documentation of progression or symptomatic deterioration, early discontinuation of treatment, or death due to any cause.
Time Frame: assessed up to 3 years post registration
Population: Eligible participants who were randomized to study arms.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Number analyzed (Participants) | 83 | 85
months | 10.8 [7.7 to 12.9] | 10.0 [7.1 to 13.5]
Statistical Analysis 1: Comparison: Arm I (Afatinib Dimaleate, Cetuximab) vs Arm II (Afatinib Dimaleate); Test type: Superiority; p = 0.95, Log Rank; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.73 to 1.39]

6. Secondary Outcome: Number of Patients With Gr 3 Through 5 Adverse Events That Are Related to Study Drugs
Description: Routine Adverse Events are reported by CTCAE4.0. For serious adverse event reporting, we updated from CTCAE4.0 to CTCAE5.0. . Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Population: Patients who received at least one dose of protocol treatment.
Measure: Number; unit: Participants
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
Number analyzed (Participants) | 78 | 85
Participants
  Abdominal pain | 1 | 0
  Acidosis | 1 | 0
  Acute kidney injury | 1 | 1
  Alanine aminotransferase increased | 1 | 1
  Alkaline phosphatase increased | 1 | 1
  Allergic reaction | 2 | 0
  Anemia | 1 | 1
  Anorexia | 0 | 1
  Aspartate aminotransferase increased | 1 | 0
  Atrial fibrillation | 0 | 1
  Back pain | 1 | 0
  Bullous dermatitis | 1 | 0
  Chills | 1 | 0
  Cough | 1 | 0
  Creatinine increased | 0 | 2
  Dehydration | 2 | 2
  Diarrhea | 12 | 17
  Dry skin | 3 | 0
  Dyspepsia | 1 | 0
  Dyspnea | 2 | 0
  Encephalopathy | 0 | 1
  Enterocolitis infectious | 0 | 1
  Fatigue | 1 | 1
  Flank pain | 1 | 0
  General disorders and admin site conditions - Other | 0 | 1
  Hypertension | 0 | 1
  Hypocalcemia | 1 | 0
  Hypokalemia | 5 | 5
  Hypomagnesemia | 1 | 0
  Hyponatremia | 0 | 1
  Hypophosphatemia | 1 | 0
  Hypotension | 1 | 0
  Hypoxia | 1 | 0
  Infections and infestations - Other, specify | 1 | 0
  Infusion related reaction | 2 | 0
  Lipase increased | 0 | 1
  Lung infection | 1 | 0
  Lymphocyte count decreased | 1 | 2
  Lymphocyte count increased | 0 | 1
  Mucositis oral | 6 | 4
  Nausea | 2 | 3
  Oral pain | 0 | 1
  Palmar-plantar erythrodysesthesia syndrome | 0 | 1
  Papulopustular rash | 2 | 0
  Paronychia | 4 | 1
  Pneumonitis | 3 | 0
  Pruritus | 3 | 1
  Rash acneiform | 21 | 2
  Rash maculo-papular | 10 | 0
  Rash pustular | 1 | 0
  Sepsis | 0 | 1
  Skin and subcutaneous tissue disorders - Other | 1 | 0
  Skin infection | 0 | 1
  Thromboembolic event | 1 | 0
  Urticaria | 1 | 0
  Vomiting | 0 | 1
  Weight loss | 1 | 0

7. Other Pre Specified Outcome: Change in Copy Number Alterations in MET, EGFR, and HER2, Analyzed Using Fluorescence in Situ Hybridization
Description: For each of these markers, a one-sample t-test (or Wilcoxon signed-rank test) will be used to test the null hypothesis that the absolute difference between the copy number after progression and the copy number in the pre-treatment specimen (or an appropriate transformation of the difference, determined after exploratory data analysis) is not equal to zero.
Time Frame: Baseline up to 3 years (after disease progression)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Change in the Ratio of Sensitizing EGFR Mutation to EGFR T790 Mutation
Description: To evaluate if EGFRs/EGFR T790M is lower at progression than in pre-treatment specimens among patients with results available for pre-treatment and progression, a one-sample t-test (or Wilcoxon signed-rank test) will be used to test the null hypothesis that the difference between the progression ratio and the pre-treatment ratio (or an appropriate transformation of the difference, determined after exploratory data analysis) is greater than zero in favor of the alternative that the difference is less than zero.
Time Frame: Baseline up to 3 years (at progression)
Reporting Status: Not Posted

9. Other Pre Specified Outcome: EGFR Immunohistochemistry H-score
Description: To evaluate the hypothesis that H-score positive status at baseline is associated with absolute difference in PFS (and OS) among patients randomized to receive afatinib dimaleate monotherapy a test of interaction will be performed at the 1-sided 20% level.
Time Frame: Baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Levels of Circulating Tumor Markers
Description: Tumor marker levels over time will be evaluated using a linear mixed model for continuous markers and using generalized estimating equations for binary markers. A landmark analysis will be used to evaluate the correlation between post-randomization biomarker values and PFS and OS (from the landmark timepoint) using a Cox proportional hazards model.
Time Frame: Up to 3 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Presence of de Novo EGFR T790M Mutation or Other Molecular Alterations
Description: To evaluate if the presence of de novo T790M mutation is associated with primary resistance to afatinib dimaleate, PFS and OS will be compared between T790M mutation positive and negative patients randomized to the afatinib dimaleate monotherapy arm using a log-rank test..
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Ratio of Sensitizing EGFR Mutation to EGFR T790 Mutation
Description: To evaluate if the ratio of EGFR sensitizing mutation to EGFR T790M mutation (EGFRs/EGFR T790M) among patients with T790M is predictive for afatinib dimaleate monotherapy, analyses will be performed in a similar fashion to the evaluation of T790M among patients with measurable T790M (which defines T790M). Cox regression will be used to assess the predictive association of the ratio in the afatinib dimaleate monotherapy arm with both OS and PFS
Time Frame: Up to 3 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Duration of treatment and follow up until death or 3 years post registration
Description: Of 168 eligible participants, 5 did not receive protocol therapy so were not assessed for AEs. Therefore only 163 participants (78 on arm 1 and 85 on arm 2) were assessed for AEs. All eligible participants were assessed for All-Cause Mortality.
Arm/Group | Arm I (Afatinib Dimaleate, Cetuximab) | Arm II (Afatinib Dimaleate)
All-Cause Mortality (participants affected / at risk) | 30/83 | 35/85
Serious Adverse Events (participants affected / at risk) | 29/78 | 30/85
Other Adverse Events (participants affected / at risk) | 78/78 | 84/85
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Afatinib Dimaleate, Cetuximab) (N=78) | Arm II (Afatinib Dimaleate) (N=85)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Lymph node pain (Blood and lymphatic system disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 7
Esophageal ulcer (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 4
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Death NOS (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Allergic reaction (Immune system disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Catheter related infection (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Infections and infestations-Other (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 2
Paronychia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 2
Skin infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Creatinine increased (Investigations) | 1 | 1
Lymphocyte count decreased (Investigations) | 1 | 0
Weight loss (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 4
Headache (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 1 | 0
Nervous system disorders-Other (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 1
Stroke (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 0
Confusion (Psychiatric disorders) | 0 | 3
Depression (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1
Hematuria (Renal and urinary disorders) | 1 | 0
Renal and urinary disorders-Other (Renal and urinary disorders) | 1 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 0
Thromboembolic event (Vascular disorders) | 5 | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Afatinib Dimaleate, Cetuximab) (N=78) | Arm II (Afatinib Dimaleate) (N=85)
Anemia (Blood and lymphatic system disorders) | 28 | 32
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 4 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 1
Cardiac disorders-Other (Cardiac disorders) | 4 | 0
Chest pain - cardiac (Cardiac disorders) | 0 | 2
Palpitations (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 4 | 6
Congenital, familial and genetic disorders - Other (Congenital, familial and genetic disorders) | 1 | 0
Ear and labyrinth disorders-Other (Ear and labyrinth disorders) | 2 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 5
External ear inflammation (Ear and labyrinth disorders) | 1 | 0
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Cushingoid (Endocrine disorders) | 0 | 1
Endocrine disorders-Other (Endocrine disorders) | 0 | 1
Blurred vision (Eye disorders) | 11 | 9
Cataract (Eye disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 13 | 7
Corneal ulcer (Eye disorders) | 1 | 0
Dry eye (Eye disorders) | 19 | 15
Eye disorders-Other (Eye disorders) | 9 | 10
Eye pain (Eye disorders) | 1 | 3
Eyelid function disorder (Eye disorders) | 1 | 0
Floaters (Eye disorders) | 0 | 1
Keratitis (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 0 | 2
Vitreous hemorrhage (Eye disorders) | 0 | 1
Watering eyes (Eye disorders) | 9 | 9
Abdominal distension (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 13 | 9
Anal hemorrhage (Gastrointestinal disorders) | 1 | 0
Bloating (Gastrointestinal disorders) | 2 | 1
Cheilitis (Gastrointestinal disorders) | 6 | 8
Constipation (Gastrointestinal disorders) | 31 | 17
Diarrhea (Gastrointestinal disorders) | 73 | 78
Dry mouth (Gastrointestinal disorders) | 10 | 14
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 8 | 8
Dysphagia (Gastrointestinal disorders) | 2 | 8
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Esophageal pain (Gastrointestinal disorders) | 1 | 0
Esophagitis (Gastrointestinal disorders) | 2 | 3
Flatulence (Gastrointestinal disorders) | 2 | 2
Gastritis (Gastrointestinal disorders) | 0 | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 8 | 8
Gastrointestinal disorders-Other (Gastrointestinal disorders) | 8 | 10
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 0
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 0 | 1
Hemorrhoids (Gastrointestinal disorders) | 3 | 2
Lip pain (Gastrointestinal disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 38 | 39
Nausea (Gastrointestinal disorders) | 44 | 34
Oral hemorrhage (Gastrointestinal disorders) | 1 | 1
Oral pain (Gastrointestinal disorders) | 4 | 2
Periodontal disease (Gastrointestinal disorders) | 1 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 1 | 4
Tooth discoloration (Gastrointestinal disorders) | 0 | 1
Toothache (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 31 | 21
Chills (General disorders) | 11 | 4
Edema face (General disorders) | 2 | 0
Edema limbs (General disorders) | 15 | 17
Fatigue (General disorders) | 58 | 49
Fever (General disorders) | 10 | 8
Flu like symptoms (General disorders) | 7 | 8
Gait disturbance (General disorders) | 1 | 2
General disorders and admin site conditions - Other (General disorders) | 11 | 9
Infusion related reaction (General disorders) | 7 | 0
Infusion site extravasation (General disorders) | 1 | 0
Irritability (General disorders) | 1 | 1
Localized edema (General disorders) | 2 | 0
Malaise (General disorders) | 1 | 1
Neck edema (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 7 | 7
Pain (General disorders) | 20 | 14
Hepatobiliary disorders-Other (Hepatobiliary disorders) | 0 | 1
Allergic reaction (Immune system disorders) | 5 | 0
Immune system disorders-Other (Immune system disorders) | 0 | 1
Bladder infection (Infections and infestations) | 0 | 2
Bronchial infection (Infections and infestations) | 3 | 2
Catheter related infection (Infections and infestations) | 0 | 1
Conjunctivitis infective (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 1
Eye infection (Infections and infestations) | 1 | 1
Infections and infestations-Other (Infections and infestations) | 11 | 17
Laryngitis (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 1 | 0
Mucosal infection (Infections and infestations) | 2 | 0
Nail infection (Infections and infestations) | 2 | 2
Otitis media (Infections and infestations) | 1 | 1
Papulopustular rash (Infections and infestations) | 7 | 5
Paronychia (Infections and infestations) | 39 | 34
Pelvic infection (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 4 | 0
Rhinitis infective (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 2 | 7
Skin infection (Infections and infestations) | 10 | 8
Tooth infection (Infections and infestations) | 0 | 2
Upper respiratory infection (Infections and infestations) | 7 | 6
Urinary tract infection (Infections and infestations) | 10 | 16
Vaginal infection (Infections and infestations) | 3 | 2
Wound infection (Infections and infestations) | 0 | 1
Bruising (Injury, poisoning and procedural complications) | 3 | 3
Burn (Injury, poisoning and procedural complications) | 0 | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 3
Injury, poison and procedural complications - Other (Injury, poisoning and procedural complications) | 2 | 2
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 21 | 24
Alkaline phosphatase increased (Investigations) | 22 | 23
Aspartate aminotransferase increased (Investigations) | 27 | 23
Blood bilirubin increased (Investigations) | 9 | 9
Cholesterol high (Investigations) | 1 | 0
Creatinine increased (Investigations) | 14 | 21
INR increased (Investigations) | 1 | 1
Investigations-Other (Investigations) | 3 | 9
Lipase increased (Investigations) | 0 | 2
Lymphocyte count decreased (Investigations) | 18 | 14
Lymphocyte count increased (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 3 | 6
Weight gain (Investigations) | 6 | 5
Weight loss (Investigations) | 22 | 29
White blood cell decreased (Investigations) | 13 | 10
Anorexia (Metabolism and nutrition disorders) | 30 | 31
Dehydration (Metabolism and nutrition disorders) | 6 | 4
Glucose intolerance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 17 | 20
Hyperkalemia (Metabolism and nutrition disorders) | 7 | 5
Hypermagnesemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 7 | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 25 | 19
Hypocalcemia (Metabolism and nutrition disorders) | 21 | 12
Hypoglycemia (Metabolism and nutrition disorders) | 4 | 3
Hypokalemia (Metabolism and nutrition disorders) | 31 | 20
Hypomagnesemia (Metabolism and nutrition disorders) | 42 | 18
Hyponatremia (Metabolism and nutrition disorders) | 12 | 18
Hypophosphatemia (Metabolism and nutrition disorders) | 4 | 2
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Arthritis (Musculoskeletal and connective tissue disorders) | 3 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 23 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 6 | 4
Buttock pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 6 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 4
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 9
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 4 | 3
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal and connective tiss disorder - Other (Musculoskeletal and connective tissue disorders) | 10 | 15
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 8
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 7 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 18
Neoplasms benign, malignant and unspecified - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 5
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Amnesia (Nervous system disorders) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 1
Concentration impairment (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 18 | 13
Dysgeusia (Nervous system disorders) | 17 | 20
Dysphasia (Nervous system disorders) | 0 | 1
Facial nerve disorder (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 23 | 22
Memory impairment (Nervous system disorders) | 7 | 3
Nervous system disorders-Other (Nervous system disorders) | 2 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Paresthesia (Nervous system disorders) | 3 | 3
Peripheral motor neuropathy (Nervous system disorders) | 1 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 9
Presyncope (Nervous system disorders) | 1 | 0
Sinus pain (Nervous system disorders) | 0 | 3
Spasticity (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 2
Agitation (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 14 | 6
Confusion (Psychiatric disorders) | 3 | 5
Depression (Psychiatric disorders) | 10 | 4
Insomnia (Psychiatric disorders) | 13 | 10
Libido decreased (Psychiatric disorders) | 1 | 0
Psychiatric disorders-Other (Psychiatric disorders) | 0 | 2
Restlessness (Psychiatric disorders) | 2 | 1
Suicide attempt (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Bladder spasm (Renal and urinary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 1
Cystitis noninfective (Renal and urinary disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 5 | 1
Proteinuria (Renal and urinary disorders) | 2 | 3
Renal and urinary disorders-Other (Renal and urinary disorders) | 4 | 3
Renal calculi (Renal and urinary disorders) | 1 | 2
Renal colic (Renal and urinary disorders) | 2 | 1
Urinary frequency (Renal and urinary disorders) | 3 | 2
Urinary tract pain (Renal and urinary disorders) | 1 | 2
Urinary urgency (Renal and urinary disorders) | 2 | 0
Irregular menstruation (Reproductive system and breast disorders) | 2 | 0
Menorrhagia (Reproductive system and breast disorders) | 2 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 3
Reproductive system and breast disorders - Other (Reproductive system and breast disorders) | 1 | 1
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal dryness (Reproductive system and breast disorders) | 0 | 2
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 16 | 9
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 36 | 36
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 | 23
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 | 20
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 13 | 8
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Resp, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11 | 12
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 13 | 13
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 48 | 37
Erythema multiforme (Skin and subcutaneous tissue disorders) | 3 | 4
Hirsutism (Skin and subcutaneous tissue disorders) | 8 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 2
Hypertrichosis (Skin and subcutaneous tissue disorders) | 2 | 2
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discoloration (Skin and subcutaneous tissue disorders) | 5 | 8
Nail loss (Skin and subcutaneous tissue disorders) | 7 | 6
Nail ridging (Skin and subcutaneous tissue disorders) | 8 | 10
Pain of skin (Skin and subcutaneous tissue disorders) | 3 | 1
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 | 9
Photosensitivity (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 32 | 26
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 62 | 50
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 36 | 32
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 2
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 34 | 21
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin induration (Skin and subcutaneous tissue disorders) | 1 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 2
Surgical and medical procedures-Other (Surgical and medical procedures) | 3 | 2
Flushing (Vascular disorders) | 2 | 1
Hot flashes (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 19 | 27
Hypotension (Vascular disorders) | 8 | 3
Lymphedema (Vascular disorders) | 0 | 1
Thromboembolic event (Vascular disorders) | 1 | 3
Vascular disorders-Other (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-07-29): https://cdn.clinicaltrials.gov/large-docs/22/NCT02438722/Prot_SAP_ICF_000.pdf